CLINICAL TRIAL: NCT06094348
Title: The Evaluation of the Effect of Piezo and Endonasal Osteotomy Methods on Postoperative Healing Process in Septorhinoplasty by the Ultrasonic Measurement of Nasal Skin Thickness
Brief Title: The Evaluation of Piezo and Endonasal Osteotomy Methods on Postoperative Healing Process in Septorhinoplasty
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Haseki Training and Research Hospital (Other)
Responsible Party: Principal Investigator, ISIL TAYLAN CEBI, principal investigator, Haseki Training and Research Hospital
Other Study IDs: Piezo vs Endonasal osteotomy
Record Dates: First submitted 2023-10-10; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Nasal Deformity, Acquired; Septum; Deviation, Congenital
Keywords: rhinoplasty; edema; piezosurgery; osteotomy
MeSH Terms: conditions — Nose Deformities, Acquired; Edema

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (4):
- Group 1A- Thick skin, endonasal osteotomy: Patients with mean nasal soft tissue envelope thickness > 4 mm undergoing classical endonasal osteotomy procedure during rhinoplasty operation
  Interventions: Procedure: Endonasal osteotomy
- Group 1B -Thick skin, piezo osteotomy: Patients with mean nasal soft tissue envelope thickness > 4 mm undergoing piezosurgery assisted osteotomy procedure during rhinoplasty operation
  Interventions: Device: Piezo assisted osteotomy
- Group 2A- Thin skin, endonasal osteotomy: Patients with mean nasal soft tissue envelope thickness <4 mm undergoing classical endonasal osteotomy procedure during rhinoplasty operation
  Interventions: Procedure: Endonasal osteotomy
- Group 2B- Thin skin, piezo osteotomy: Patients with mean nasal soft tissue envelope thickness < 4 mm undergoing piezosurgery assisted osteotomy procedure during rhinoplasty operation
  Interventions: Device: Piezo assisted osteotomy

INTERVENTIONS:
Procedure: Endonasal osteotomy — Patients will undergo median-oblique and lateral osteotomy, with conventional 2 mm guarded, straight osteotome.
  Groups: Group 1A- Thick skin, endonasal osteotomy; Group 2A- Thin skin, endonasal osteotomy
Device: Piezo assisted osteotomy — Piezo is a system for cutting bone with micrometric ultrasonic piezoelectric vibrations, with varying frequency and cutting energy. The device consists of a platform with a powerful piezoelectric hand piece and employs a functional frequency between 25-29 kHz. The device is fitted with a cooling irrigation system with a 0-60 cc/min variable sterile solution flow. Specific inserts and scalpels act in a linear vibration pattern, with a spatial range between 60 and 210 microns, moved by an ultrasonic power that exceeds 5 watts, reaching up to 16 watts.
  Groups: Group 1B -Thick skin, piezo osteotomy; Group 2B- Thin skin, piezo osteotomy

SUMMARY:
The goal of this observational study is to compare the effect of Piezo and endonasal osteotomy techniques on the healing process of patients undergoing septorhinoplasty surgery. The main question[s] it aims to answer are:

* In which osteotomy technique the edema is lesser?
* Which osteotomy technique is better for thick vs thin skinned patients ? In which osteotomy technique the healing process is faster?

Participants will be asked to have an ultrasonic measurement of the nasal dorsum preoperatively and at the first, third and tenth months postoperatively.

Researchers will compare the thick and thin skinned patients to detect which osteotomy technique is superior in the healing process ( lesser edema and faster healing due to skin thickness measurements)

DETAILED DESCRIPTION:
The goal of this observational study is to compare the effect of Piezo and endonasal osteotomy techniques on the healing process of patients undergoing septorhinoplasty surgery. The main question[s] it aims to answer are:

* In which osteotomy technique the edema is lesser?
* Which osteotomy technique is better for thick vs thin skinned patients ? In which osteotomy technique the healing process is faster?

18-65 years old males or females with nasal septum and/or nasal pyramid deviation and external nasal deformities who are willing to undergo open rhinoplasty procedure will be included in the study. Patients who have a history of previous rhinoplasty/septorhinoplasty procedure, abnormal coagulation parameters (prothrombin time, partial thromboplastin time, bleeding/coagulation time), use of anticoagulant drugs, chronic / inflammatory skin disease and/or chronic skin allergies, systemic diseases (hypertension, diabetes mellitus, bronchial asthma), nasal beautification procedures such as dermal fillings, using oral and/or topical (nasal skin) corticosteroids in three months preoperatively will be excluded.

Participants will be asked to have an ultrasonic measurement of the nasal dorsum preoperatively and at the first, third and tenth months postoperatively.

Researchers will compare the thick and thin skinned patients to detect which osteotomy technique is superior in the healing process ( lesser edema and faster healing due to skin thickness measurements).

ELIGIBILITY:
Inclusion Criteria:

* nasal respiratory dysfunction with the deviation of nasal septum and/or the nasal pyramid

Exclusion Criteria:

* previous rhinoplasty/septorhinoplasty procedure
* patients with abnormal coagulation parameters (prothrombin time, partial thromboplastin time, bleeding/coagulation time)
* use of anticoagulant drugs
* chronic / inflammatory skin disease and/or chronic skin allergies
* presence of systemic diseases (hypertension, diabetes mellitus, bronchial asthma)
* nasal beautification procedures such as dermal fillings
* use of oral and/or topical (nasal skin) corticosteroids in three months preoperatively

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 18-65 year, males or females with nasal septum and/or nasal pyramid deviation and external nasal deformities who are willing to undergo open rhinoplasty procedure.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-05-19 (Actual); Primary Completion 2024-04-19 (Estimated); Study Completion 2024-04-19 (Estimated)

PRIMARY OUTCOMES:
the mean nasal soft tissue envelope thickness measurements of rhinoplasty patients at postoperative 10th month | 10 months
  the mean nasal soft tissue envelope thickness measurements of rhinoplasty patients at postoperative 10 th month will be done by ultrasonography at four anatomic locations; these locations are nasion, rhinion, supratip and tip

CONTACTS AND LOCATIONS:
Overall Officials: Isil Taylan Cebi, M.D, Principal Investigator — Haseki Training and Research Hospiral
Locations (1):
- Haseki Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gode S, Ozturk A, Kismali E, Berber V, Turhal G. The Effect of Platelet-Rich Fibrin on Nasal Skin Thickness in Rhinoplasty. Facial Plast Surg. 2019 Aug;35(4):400-403. doi: 10.1055/s-0039-1693436. Epub 2019 Jul 15. PMID 31307096
- [Background] Erdur ZB, Oktem F, Inci E, Yener HM, Ustundag A. Effect of Nasal Soft-Tissue Envelope Thickness on Postoperative Healing Process Following Rhinoplasty. J Craniofac Surg. 2021 Sep 1;32(6):2193-2197. doi: 10.1097/SCS.0000000000007697. PMID 33867511
- [Background] Stenner M, Koopmann M, Rudack C. Measuring the nose in septorhinoplasty patients: ultrasonographic standard values and clinical correlations. Eur Arch Otorhinolaryngol. 2017 Feb;274(2):855-860. doi: 10.1007/s00405-016-4296-7. Epub 2016 Sep 15. PMID 27628964
- [Background] Tsikopoulos A, Tsikopoulos K, Doxani C, Vagdatli E, Meroni G, Skoulakis C, Stefanidis I, Zintzaras E. Piezoelectric or Conventional Osteotomy in Rhinoplasty? A Systematic Review and Meta-Analysis of Clinical Outcomes. ORL J Otorhinolaryngol Relat Spec. 2020;82(4):216-234. doi: 10.1159/000506707. Epub 2020 Apr 22. PMID 32320977
- [Background] Kurt Yazar S, Serin M, Rakici IT, Sirvan SS, Irmak F, Yazar M. Comparison of piezosurgery, percutaneous osteotomy, and endonasal continuous osteotomy techniques with a caprine skull model. J Plast Reconstr Aesthet Surg. 2019 Jan;72(1):107-113. doi: 10.1016/j.bjps.2018.08.025. Epub 2018 Sep 4. PMID 30243555